CLINICAL TRIAL: NCT05002803
Title: The Development and Validation of the Arabic Otago Exercise Program: A Feasibility Controlled Study
Brief Title: The Development and Validation of the Arabic Otago Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Alia A. Alghwiri, Professor, University of Jordan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/134
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Older Adults
Keywords: Otago Exercise Program; Falls; Older adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program (Experimental): Older adults will receive the Arabic Otago Exercise Program for 8 weeks plus health awareness videos.
  Interventions: Other: Otago Exercise Program
- Control group (No Intervention): Older adults will receive only health awareness videos every 2 weeks.

INTERVENTIONS:
Other: Otago Exercise Program — A Home-based Exercise Program to improve strength and balance and prevent falls.
  Arms: Otago Exercise Program

SUMMARY:
Falls are common in older adults and may lead to disability or even death. Therefore, exercise programs that focus on preventing falls by improving strength and balance are important to investigate in older adults. One of the home-based exercise programs that was found effective in reducing the risk of falling and the rate of subsequent falls in older adults is the Otago exercise program (OEP). The OEP is an individualized home based retraining program that works mainly on balance and lower extremity strength through several progressive resistive exercises.

The OEP is available in English language since late 1990. However, its use in the Arabic-speaking countries is limited due to the language barrier. Therefore, translating such a program to the Arabic language would facilitate its use among Arabic-speaking older adults.

Therefore, this study aims:

* To translate the Otago Exercise Program (OEP) into the Arabic language.
* To assess the feasibility of the Arabic OEP in a pilot sample of Arabic-speaking older adults.

DETAILED DESCRIPTION:
* Research ethics: This study got the ethics approval from the IRB at Jordan University Hospital at University of Jordan. A consent form that contains the study procedures will be prepared and signed from all participants. To insure the privacy of participants, every older adult will be assigned a study identification number. All results will be stored in a locked cabinet/computer only accessible by the researchers.
* Participants: Data will be collected prospectively from older adults in Jordan. Older adults will be approached to complete the program via Jordan University Hospital, community based organizations (e.g. Help-Age International Jordan) and social media platforms such as Facebook and WhatsApp.

Design:

Phase 1: Translation and cultural adaptation of the Otago Exercise Program (OEP) into the Arabic language.

* The permission of translating the program will be granted from its developers.
* English version of the program will be translated into the Arabic language in accordance with the World Health Organization (WHO) forward/backward translation protocol (https://www.who.int/substance_abuse/research_tools/translation/en/ ).
* An Arabic booklet of the OEP will be prepared.

Phase 2: Assessing feasibility of the OEP on a pilot sample of Arabic-speaking older adults using a focus group and a pilot Trial.

* The Arabic version of the OEP will be sent to an expert panel for review. Suggested changes will be considered and made.
* The Arabic version of the OEP will be sent to 2 groups that consist of 5 older adults each. They will be given sufficient time to go through the exercise manual before being invited to a focus group meeting to discuss the Arabic wording and feasibility of the Arabic version of the OEP.
* A topic guide will be prepared to assess the feasibility and user-friendliness of the Arabic OEP manual.
* The meeting will be recorded after taking their permission and the recording will be transcribed and analyzed.
* If there are major changes to the program, the experts will meet to make the appropriate changes and another focus group will be conducted.
* The final version of the Arabic OEP will be implemented for 8 weeks on a pilot sample of Arabic speaking older adults using a controlled design with 10 older adults in the treatment group and 10 older adults in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are 60 years of age and older.
* Who can read and write in Arabic language.
* Who are able to walk outdoors with no more support than a single point cane.

Exclusion Criteria:

* Who have a serious orthopedic condition (e.g., recent lower limb surgery, severe arthritis of a lower limb) or major neurological disorder (e.g., stroke with unilateral or bilateral paresis, Parkinson disease or multiple sclerosis) that could restrict functional mobility.
* Who are unable to comprehend study information and consent processes due to any illness including dementia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Falls in the previous 12 months | Previous 12 months
  Incidence of Falls and Falls Circumstances in the previous 12 months
Incidence of falls during the treatment period (8 weeks) | Immediately post intervention.
  Incidence of falls during the treatment period (previous 2 months) to assess the effect of the intervention on the incidence of falls.

SECONDARY OUTCOMES:
Fear of Falling (using the Falls Efficacy Scale-International) | Immediately post intervention.
  The effect of the intervention on fear of falling. The total score ranges between 16 and 64 with a higher score indicates greater fear of falling (worse).
Balance (using Chair balance test and Four test balance scale) | Immediately post intervention.
  The effect of the intervention on balance. The time taken to conduct these balance tasks are timed using a stopwatch. The longer the time taken by the participant to perform the tasks, the worse the balance. There is no minimum or maximum scores for these tests.
Mobility (using Timed-Up and go) | Immediately post intervention.
  The effect of the intervention on mobility. This assessments of mobility is timed out using a stopwatch.
Grip strength (using a hand held dynamometer) | Immediately post intervention.
  The effect of the intervention on grip strength. The strength of Hand grip muscle will be assessed using a dynamometer in kilograms.
The Quality of Life (using Medical Outcomes Study Short Form 12) | Immediately post intervention.
  The effect of the intervention on Quality of Life. The total score ranges between 0% to 100% with higher score indicates a better quality of life (better).
The severity of Anxiety and Depression (using Hospital Anxiety and Depression Scale) | Immediately post intervention.
  The effect of the intervention on the severity of Anxiety and Depression. The total score for each subscale of the HADS ranges from 0 to 21 with higher score indicates more severe anxiety or depression (worse).
Pain (using pain rating scale) | Immediately post intervention.
  The effect of the intervention on pain. The total score of PRS ranges between 0 to 10 with higher score indicates more pain and interference with discomfort (worse).
The severity of fatigue (using the Modified Fatigue Impact Scale) | Immediately post intervention.
  The effect of the intervention on fatigue. The total score of MFIS ranges between 0 to 84 with higher score indicates higher impact of fatigue on on daily functioning (worse).

CONTACTS AND LOCATIONS:
Overall Officials: Alia A. Alghwiri, PhD, Principal Investigator — University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No